CLINICAL TRIAL: NCT01754064
Title: St. Jude Medical Product Longevity and Performance (SCORE) Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 40007941/F
Record Dates: First submitted 2012-12-13; First posted 2012-12-21 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Bradycardia; Tachycardia; Heart Disease
Keywords: Bradycardia; Tachycardia; Arrhythmia; ICD; pacemaker; pacing lead
MeSH Terms: conditions — Bradycardia; Tachycardia; Heart Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Rhythm Management device: Implanted with implantable defibrillator or pacemaker system
  Interventions: Device: Cardiac Rhythm Management device

INTERVENTIONS:
Device: Cardiac Rhythm Management device

SUMMARY:
SCORE is an active, prospective, non-randomized, multi-center outcome-oriented registry of patients implanted with St Jude Medical (SJM) market-released cardiac rhythm management (CRM) products. This registry will be conducted in the United States (US).

The primary purpose of the registry is to evaluate and publish acute and long-term performance of market-released SJM CRM products by analyzing product survival probabilities. Product status and any related adverse events will be collected to measure survival probabilities.

ELIGIBILITY:
Enrollment Criteria:

* Patient has a standard indication for a CRM implantable device.
* Patient is implanted with at least one new market-released SJM CRM product from a list provided by SJM (e.g pacemaker, ICD, CRT-D, CRT-P, pacing/sensing lead, defibrillation lead) within the last 90 days.
* Complete system implant information (e.g. model, serial number, location) is available at enrollment.
* Any product-related adverse event information at implant is available at enrollment.
* Patient or appropriate legal guardian is willing to provide authorization for registry participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient indicated for a cardiac rhythm management (CRM) product like ICD, pacemaker, CRT-D, CRT-P, leads, etc. would be eligible for participation in the study.
Sampling Method: Probability Sample
Enrollment: 10957 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Event Free Survival | 5 year average

CONTACTS AND LOCATIONS:
Overall Officials: Grant Kim, Study Director — Abbott Medical Devices
Locations (80):
- United States (80):
  - Heart Center Research, LLC., Huntsville, Alabama
  - Cardiology Associates of Mobile, Inc., Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Arizona Cardiovascular Research Center, Phoenix, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Pima Heart Physicians, PC, Tucson, Arizona
  - Northwest Cardiology, Springdale, Arkansas
  - Raymond Schaerf, MD, Burbank, California
  - California Heart Medical Associates, Fresno, California
  - Glendale Memorial Hospital and Medical Center, Glendale, California
  - Jeffrey Goodman MD, Los Angeles, California
  - Cardiac Rhythm Specialists, Inc., Reseda, California
  - Truong Duong MD, Riverside, California
  - Mercy Medical Group - Cardiology, Sacramento, California
  - Pacific Heart Institute, Santa Monica, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Michael Pittaro MD, New Canaan, Connecticut
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Cardiac Arrhythmia Services, Boca Raton, Florida
  - Shands Jacksonville, Jacksonville, Florida
  - Jorge Diaz, M.D., P.A., Lake Mary, Florida
  - Naples Heart Rhythm Specialists, PA, Naples, Florida
  - Central Florida Heart Center, Ocala, Florida
  - Cardiology Consultants - Baptist Campus, Pensacola, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Heart Institute - Buckhead Location, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Harbin Clinic Southeastern Cardiovascular Institute, Rome, Georgia
  - North Shore Cardiology, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Parkview Research Center, Fort Wayne, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Mid-America Cardiology Associates, PC, Kansas City, Kansas
  - King's Daughters Medical Center, Ashland, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Cardiac Associates PC, Rockville, Maryland
  - Pioneer Valley Cardiology, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Thoracic Cardio Healthcare Found. (aka Sparrow Clinical Research Institute), Lansing, Michigan
  - Ascension St. Mary's Research Institute, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Renown Institute for Heart and Vascular Health, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Morristown Memorial Hospital (Atlantic Health System), Morristown, New Jersey
  - New Jersey Cardiology Associates, West Orange, New Jersey
  - Trinity Medical WNY, PC, Buffalo, New York
  - Manhattan Cardiac Arrhythmia Consultants, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Westfall Cardiology LLP, Rochester, New York
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Allegheny Singer Research Institute, Pittsburgh, Pennsylvania
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Lexington Cardiology, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Apex Cardiology, Jackson, Tennessee
  - Memphis Cardiac Care Center, Memphis, Tennessee
  - The Heart Group, PLLC, Nashville, Tennessee
  - Vanderbilt Page-Campbell Heart Institute, Nashville, Tennessee
  - Dallas Heart Group, Dallas, Texas
  - Cardiovascular Association, P.L.L.C., Humble, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Medicine School of University Health Care, Salt Lake City, Utah
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Cardiovascular Associates of Virginia, Midlothian, Virginia
  - Eastside Cardiology Associates, Kirkland, Washington
  - Kootenai Heart Clinics, Spokane, Washington
  - Dr. Edmundo Figueroa, MD, Charleston, West Virginia
  - Cardiac & Vascular of Monongalia General Hospital, Morgantown, West Virginia
  - Dean Foundation, Madison, Wisconsin